CLINICAL TRIAL: NCT00261482
Title: An Open Label, Multicentre Study of the EVRA (Norelgestromin + Ethinyl Estradiol) Transdermal Contraceptive Patch in Europe: Evaluation of Women's Experience With EVRA� and Comparison With Previously Used Methods of Contraception.
Brief Title: Evaluation of Women's Experience With EVRA (Norelgestromin + Ethinyl Estradiol) Transdermal Contraceptive Patch Compared With Previous Methods of Contraception.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002905
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Contraception; Female Contraception
Keywords: contraception; female contraception; hormonal contraception; transdermal contraception; EVRA; estrogen; progestin; ethinyl estradiol; norelgestromin
MeSH Terms: interventions — norelgestromin; Ethinyl Estradiol

INTERVENTIONS:
Drug: norelgestromin + ethinyl estradiol

SUMMARY:
The purpose of the study is to evaluate user experience with the EVRAÂ® Contraceptive Transdermal Patch; specifically, user satisfaction with the EVRAÂ® Patch, and if applicable, user preference of the EVRAÂ® Patch compared with the previous method of contraception. The study also evaluates contraceptive efficacy, safety and user compliance.

DETAILED DESCRIPTION:
EVRA is the first transdermal contraceptive patch to receive approval by Health Canada and Marketing Authorization throughout the European Union. This is an open-label, single-arm, multicenter clinical study with a treatment duration of 24 weeks (6 treatment cycles of 4 weeks). Four clinic visits are scheduled: a screening Visit 1, in which subjects are asked to complete a set of questions about satisfaction with the current method of contraception, and questions about overall health status. Visits 2, 3, and 4 follow after Cycles 1, 3, and 6, respectively of EVRA treatment. At Visits 3 and 4, the subjects are asked to answer questions about satisfaction with EVRA, and about overall health status. At Visit 4 (final study visit) the subjects are asked to compare EVRA with previously used contraceptive methods. Compliance is assessed at all visits by returned boxes of study medication and a review of Diary Cards where subjects recorded the dates and sites of patch application, and details of any patch detachment. The study will generate the first large-scale, European dataset on women's experience with EVRA, including satisfaction, safety, efficacy, and compliance. These data will be compared with subjects' experience with previously used methods of contraception. Each EVRA patch, containing 6 mg NGMN and 600 ug EE, and delivering 150 microgram NGMN and 20 ug EE over 24 hours for 7 days, is worn for 1 week and replaced for 3 consecutive weeks. The fourth week is patch-free. Subjects can wear EVRA on 1 of 4 areas: buttock, abdomen, upper torso, or upper arm.

ELIGIBILITY:
Inclusion Criteria:

* Regular menstrual cycles
* sexually active and at risk of pregnancy
* nonpregnant
* normal Pap smear

Exclusion Criteria:

* Presently have or at risk of venous thrombosis or arterial thrombosis
* migraines with focal aura
* severe hypertension
* diabetes mellitus
* hereditary dyslipoproteinemia
* carcinoma of breast, endometrium or other estrogen-dependent neoplasia
* substance abuse
* skin conditions
* concurrent use of hormone-containing medication
* smoking women over 35 years of age.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 778 (Actual)
Dates: Start 2003-07; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Level of satisfaction with EVRA after 3 and 6 cycles of use. Comparisons are made between EVRA satisfaction level and that with the previous primary contraceptive method.

SECONDARY OUTCOMES:
Efficacy is determined using the Pearl Index and the life table analysis (gross cumulative probability of pregnancy). Safety is evaluated throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.